CLINICAL TRIAL: NCT05787067
Title: The Effect of Health Belief Model-Based Mobile Online Training Applied to Patients With Diabetes on Insulin Therapy
Brief Title: The Effect of Mobile Online Training Applied to Patients With Diabetes on Insulin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Büşra Ceren DEMİREL YILDIZ, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BÜŞRA TEZ
Record Dates: First submitted 2023-02-22; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes; web-based mobile training; insulin therapy; insulin self-management; insulin injection skill; health belief model
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The web-based "Insulin Guide" mobile application prepared by the researcher was installed on the phones of the intervention group participants. They were asked to use this application for three months, at least three hours a week. Participants were followed up through the application. Participants who did not use the application were informed by SMS or phone and asked to use the application. Participants who did not use the application were excluded from the study. At the end of three months, the participants in the intervention groups were invited to the Endocrinology and Metabolic Diseases Outpatient Clinic for a post-test. Both groups were asked to practice again on the insulin injection model. Whether the application was correct, incomplete, or incorrect was recorded on the observation form by the diabetes nurse.
  Interventions: Behavioral: Health Belief Model-Based Mobile Online Training
- control group (No Intervention): Control group participants were invited to the Endocrinology and Metabolic Diseases Polyclinic for the pre-test. They were asked to administer insulin injections using an insulin injection model. Whether the application was correct, incomplete or incorrect was recorded in the observation form by the diabetes nurse. No intervention was made to the participants. At the end of three months, the participants in the control group were invited to the Endocrinology and Metabolic Diseases Polyclinic for the final test. And they were asked to repeat the insulin injection model. Whether the application was correct, incomplete or incorrect was recorded in the observation form by the diabetes nurse.

INTERVENTIONS:
Behavioral: Health Belief Model-Based Mobile Online Training — Health Belief Model-Based Mobile Online Training
  Arms: Intervention group

SUMMARY:
This study aims to investigate the effect of health belief model-based mobile online training applied to patients with diabetes on insulin therapy.

DETAILED DESCRIPTION:
Intervention and control group participants were invited to the Endocrinology and Metabolic Diseases Outpatient Clinic for a pre-test. n addition, each group was given insulin injection practice training using an insulin injection model. Whether the application was correct, incomplete, or incorrect was recorded on the observation form by the diabetes nurse. The web-based "Insulin Guide" mobile application prepared by the researcher was installed on the phones of the intervention group participants. They were asked to use this application for three months, at least three hours a week. Participants were followed up through the application. Participants who did not use the application were informed by SMS or phone and asked to use the application. Participants who did not use the application were excluded from the study. No intervention was made for the control group participants. At the end of three months, the participants in the intervention and control groups were invited to the Endocrinology and Metabolic Diseases Outpatient Clinic for a post-test. Both groups were asked to practice again on the insulin injection model. Whether the application was correct, incomplete, or incorrect was recorded on the observation form by the diabetes nurse.

ELIGIBILITY:
Research Inclusion Criteria

* Type 1 DM
* Type 2 DM (Diagnosed at least six months ago)
* Patients receiving insulin therapy
* Patients in the 18-65 age group
* Literate patients
* Patients, or patients with a relative, who has an electronic device such as a smartphone, computer, etc. that can connect to the Internet.
* Patients who have no psychiatric illness or communication barrier (visual, auditory, and speech disability)
* Individuals who agreed to participate in the research.

Research Exclusion Criteria

* Patients who receive treatment with oral anti-DM only
* Patients who use an insulin pump
* Patients who quit the training.
* Patients who had a change in treatment
* Patients who traveled to a place that cannot provide an Internet connection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of Participants' Metabolic Variables (Body Mass Index (BMI) | Three months
  The metabolic variables (Body Mass Index) of the individuals in the experimental and control groups were taken from hospital records and evaluated. With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, the BMI values of individuals in both the experimental and control groups were re-evaluated from the hospital records.
Evaluation of Participants' Metabolic Variables ( Fasting Blood Sugar (FBS)) | Three months
  The metabolic variables (Fasting Blood Sugar) of the individuals in the experimental and control groups were evaluated by taking them from the hospital records. With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, the FBC values of individuals in both the experimental and control groups were re-evaluated from the hospital records.
Evaluation of Participants' Metabolic Variables (High Density Lipoprotein (HDL)) | Three months
  The metabolic variables (High Density Lipoprotein) of the individuals in the experimental and control groups were evaluated from hospital records. With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, HDL values of individuals in both the experimental and control groups were re-evaluated from hospital records.
Evaluation of Participants' Metabolic Variables (Low Density Lipoprotein (LDL)) | Three months
  The metabolic variables (Low Density Lipoprotein) of the individuals in the experimental and control groups were evaluated from hospital records. With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, the LDL values of individuals in both the experimental and control groups were re-evaluated from the hospital records.
Evaluation of Participants' Metabolic Variables (HgA1C) | Three months
  HgA1C, one of the metabolic variables of the individuals in the experimental and control groups, was taken from hospital records and evaluated. With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, HgA1C values of individuals in both the experimental and control groups were re-evaluated from hospital records.
Evaluation of Participants' Self-Management of Insulin Therapy | Three months
  Insulin therapy self-management of individuals in the experimental and control groups was evaluated with the "Insulin Therapy Self-Management Scale". With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, the insulin therapy self-management of individuals in both the experimental and control groups was re-evaluated with the "Insulin Therapy Self-Management Scale". "Insulin Therapy Self-Management Scale" is a scale used to evaluate the knowledge-skill levels and positive-negative attitudes of individuals with diabetes towards insulin therapy. The increase in the scores obtained in all sub-dimensions indicates that the self-management levels in that dimension increase.
Evaluation of Participants' Health Belief Attitudes and Behaviors | Three months
  The health belief attitudes and behaviors of the individuals in the experimental and control groups were evaluated with the "Health Belief Model Scale". With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, the health belief attitudes and behaviors of individuals in both the experimental and control groups were re-evaluated using the "Health Belief Model Scale". The scale used to evaluate the health belief attitudes and health behaviors of individuals with diabetes consists of a total of 33 items. If the score obtained from the scale is four and above, it indicates positive health belief, and if it is less than four, it indicates negative health belief.
Evaluation of Participants' Insulin Injection Administration Skill Levels | Three months
  The insulin injection application skill levels of the individuals in the experimental and control groups were evaluated with the "Insulin Injection Skill Observation Form" prepared by the researcher in line with the literature. With the developed web-based mobile "Insulin Guide" application, the experimental group was trained for three months. No intervention was made in the control group. Three months later, the insulin injection skill levels of both the experimental and control groups were re-evaluated with the "Insulin Injection Skill Observation Form". "Insulin Injection Skill Observation Form" was developed with the aim of objectively evaluating insulin injection application performance. It consists of 21 items in total. If the patient did the application wrong, he/she gets 0 points, if he/she did it incompletely, he/she gets 1 point, and if he/she did it completely, he/she gets 2 points. The higher the average score, the higher will be their insulin injection skill level.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Universty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No